CLINICAL TRIAL: NCT03173469
Title: The Role of Preoperative Breast Magnetic Resonance Imaging for Surgical Decision in Patients Undergoing Therapeutic Mammoplasty
Brief Title: Preoperative Breast Magnetic Resonance Imaging for Patients Undergoing Mammoplasty
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, A maher, Principle investigator, Assiut University
Other Study IDs: MRIbreast
Record Dates: First submitted 2017-05-30; First posted 2017-06-01 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: magnetic resonance imaging of breast — all patients will undergo preoperative MRI

SUMMARY:
all female with operable breast cancer seeking health care at general surgery department Assiut university hospitals,and decision of therapeutic mammoplasty was taken depending on clinical examination, findings on mammography and sonography, will undergo MRI breast, and see if MRI finding will change decision of the surgery.

DETAILED DESCRIPTION:
* Study Setting: Assiut university hospital, general surgery department (C unit )
* Study subjects: all female with operable breast cancer seeking health care at general surgery department and decision of therapeutic mammoplasty was taken depending on clinical examination, findings on mammography and sonography.

The size, number, and location of breast cancer lesions were identified on US and mammography.

Also size, number, location, pattern of enhancement and presence or absence of intraductal component will be evaluated by preoperative MRI.

The surgical plane will be decided based on US and mammography findings. The final decision will be based on MRI findings. When the initial surgical decision was the same as final decision the patient will be assigned to the unchanged group.

However, if the final decision differed from the initial surgical decision the patient will be assigned to the changed group.

ELIGIBILITY:
Inclusion Criteria:

* Female patient with operable breast cancer (stage 1 and 2 ) Patient meet the criteria of therapeutic mammoplasty

Exclusion Criteria:

* Inoperable breast cancer (stage 3 and 4) Breast cancer size > 4 cm in diameter Previous radiotherapy Local recurrence after previous breast conservation surgery Male breast cancer

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: All female with operable breast cancer who candidate fot therapeutic mammoplasty,Sample size was calculated using G power, it is 40 patients.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-07-15 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-08-15 (Actual)

PRIMARY OUTCOMES:
percentage of patients whom MRI finding that will change the decision of surgery | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No